CLINICAL TRIAL: NCT02076256
Title: The Influence of Helping Relationships From Significant Others on Healthy Lifestyle and Quality of Life Among Patients With Chronic Kidney Disease: A Longitudinal Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng Kung University (Other)
Collaborators: National Cheng-Kung University Hospital (Other); E-DA Hospital (Other)
Responsible Party: Principal Investigator, Miaofen Yen, PhD, RN, FAAN, National Cheng Kung University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: NSC102-2314-B-006-013-MY3
Record Dates: First submitted 2014-02-21; First posted 2014-03-03 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Kidney Diseases
Keywords: helping relationships, healthy lifestyle, quality of life
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention)
- The helping relationships intervention program (Experimental): The helping relationships intervention program will be implemented on the experimental group. And the control group will be provided with routine nursing care. Data will be collected at baseline, the sixth and the ninth month of the third year of study. Data will be analyzed using generalized estimating equation measures to evaluate the effect of the intervention program.
  Interventions: Behavioral: The helping relationships intervention program

INTERVENTIONS:
Behavioral: The helping relationships intervention program
  Arms: The helping relationships intervention program

SUMMARY:
Helping relationships from significant others may assist patients with chronic kidney diseases to exercise health behaviors. Patients will adhere on the suggestions from medical staff and perform health lifestyle to maintain healthy behavior. The progress of the disease may be delayed.

The research is a 3-year study to explore the influence of helping relationships on healthy behaviors among patients with chronic kidney disease. Building on the findings from the past three years study and the literature on trans-theoretical Model, helping relationships will be articulated. A helping relation intervention will be applied to evaluate its effect on healthy lifestyle and quality of life.

The first year study will be a survey design. An instrument to measure the helping relationship will be established and tested. Total of 200 participants will be recruited to test the reliability and validity of the instrument. After evaluating the psychometric properties of the instrument, items may be revised according to the results. The second year of research will be a cross-section study. Of 250 subjects will be recruited to explore the correlations between helping relationships, healthy life styles, and quality of life. Data will be analyzed using hierarchical linear regression. In the third year, an experimental design will be applied to test the effect of a helping relationship intervention. One hundred and twenty subjects will be recruited and randomly assigned to the experimental and the control group for 60 subjects in each group. The helping relationships intervention program will be implemented on the experimental group. And the control group will be provided with routine nursing care. Data will be collected at baseline, the sixth and the ninth month of the third year of study. Data will be analyzed using generalized estimating equation measures to evaluate the effect of the intervention program.

ELIGIBILITY:
Inclusion Criteria:

* 20 years and older
* diagnosed with chronic kidney disease stage 1 to 4 or GFR≧30ml/min/1.73m2
* patients who has significant others
* patients who can speak Mandarin or Taiwanese

Exclusion criteria:

* Patient who limited to exercise

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2013-08; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Helping Relationship Scale | First year
Health Promotion Lifestyle Profile | First year
  Health promotion was measured by 52 item health promotion lifestyle profileⅡ ( HPLP-II).
World Health Organization Quality of Life (WHOQOL-BREF) with the Short-Form 36 (SF-36) | First year
  The study will use WHOQOL-BREF to measure the outcome.
International Physical Activity Questionnaire Taiwan Version | First year
  The study will use International Physical Activity Questionnaire (IPAQ) Taiwan version to measure the outcome.
Helping Relationship Scale | Second year
Health Promotion Lifestyle Profile | Second year
  Health promotion was measured by 52 item health promotion lifestyle profileⅡ ( HPLP-II).
World Health Organization Quality of Life (WHOQOL-BREF) with the Short-Form 36 (SF-36) | Second year
  The study will use WHOQOL-BREF to measure the outcome.
International Physical Activity Questionnaire Taiwan Version | Second year
  The study will use International Physical Activity Questionnaire (IPAQ) Taiwan version to measure the outcome.
Helping Relationship Scale | The third year
Health Promotion Lifestyle Profile | The third year
  Health promotion was measured by 52 item health promotion lifestyle profileⅡ ( HPLP-II).
World Health Organization Quality of Life (WHOQOL-BREF) with the Short-Form 36 (SF-36) | The third year
  The study will use WHOQOL-BREF to measure the outcome.
International Physical Activity Questionnaire Taiwan Version | The third year
  The study will use International Physical Activity Questionnaire (IPAQ) Taiwan version to measure the outcome.
body weight | six months
Waist to Hip Ratio | six months

CONTACTS AND LOCATIONS:
Overall Officials: Miaofen Yen, Principal Investigator — National Cheng Kung University
Locations (1):
- National Cheng Kung University, Tainan, Taiwan